CLINICAL TRIAL: NCT00917462
Title: Phase II Trial of Sorafenib for Patients With Metastatic or Recurrent Esophageal and Gastroesophageal Junction Cancer
Brief Title: Sorafenib for Patients With Metastatic or Recurrent Esophageal and Gastroesophageal Junction Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Collaborators: Bayer (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 09-016
Record Dates: First submitted 2009-06-05; First posted 2009-06-10 (Estimated); Results first posted 2019-03-13 (Actual); Last update posted 2019-03-27 (Actual); Status verified 2018-08

CONDITIONS: Esophageal Cancer; Gastroesophageal Junction Cancer
Keywords: ESOPHAGUS; BAY 43-9006 (SORAFENIB); 09-016; Nexavar®.
MeSH Terms: conditions — Esophageal Neoplasms | interventions — Sorafenib

ARMS (1):
- Sorafenib (Experimental): Sorafenib for patients with metastatic or recurrent esophageal and gastroesophageal junction cancer.
  Interventions: Drug: Sorafenib, administered orally; Procedure: CT/MRI

INTERVENTIONS:
Drug: Sorafenib, administered orally — Sorafenib 400 mg twice daily administered continuously. Patients will continue on treatment until progression of disease. Each cycle consists of 28 days. The cycle start date will coincide with the physician visit date. Because of the potential need for physician visit scheduling to vary (due to both physician and patient issues), to avoid violation of, and deviation from, the protocol, these visits may vary by up to one to fourteen (1-14) days. A study diary will be completed by patients to ensure compliance with the study drug.
Procedure: CT/MRI — A CT (computerized tomography) or MRI (magnetic resonance imaging) scan of the chest and abdomen will be obtained at baseline, after the first four weeks of therapy, at eight weeks, and then every eight weeks there afterwith a scheduling window of up to one to fourteen (1-14) days. The same imaging modality performed at baseline (CT or MRI) will be repeated at subsequent imaging.

SUMMARY:
Sorafenib is a drug being studied for the treatment of cancer. Sorafenib has been shown to block certain proteins on the surface of some cancer cells called "growth factor receptors." Blocking these growth factor receptors can slow or stop cancer cell growth.

Sorafenib is also known as Nexavar®. It has been studied in other types of cancers, including kidney cancer, and has been approved by the Food and Drug Administration (FDA) for treating advanced kidney cancer. Because it is not approved by the FDA for treating esophageal cancer, it is considered an experimental treatment.

The purpose of this study is to determine what effects sorafenib has on advanced esophageal cancer. These effects include whether sorafenib can shrink the tumor or slow down its growth and what side effects sorafenib will have on the tumor.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have histologically proven or cytologically confirmed esophageal cancer (squamous cell carcinoma or adenocarcinoma) or adenocarcinoma of the gastroesophageal (GE) junction documented at MSKCC.
* Metastatic disease measurable on a CT or MRI scan. Locally recurrent disease that is not amenable to potentially curative surgery or radiation therapy is also allowed. Lesions must be ≥ 10 mm in size. The primary tumor is not considered measurable disease. Recurrent or metastatic lesions within a prior radiation field are acceptable as long as disease has progressed in the radiation field by RECIST criteria. The same imaging modality performed at baseline (CT or MRI) will be repeated at subsequent imaging.
* Patients are allowed to have a maximum of two prior chemotherapy regimens for metastatic disease. Patients are allowed to have a maximum of three prior regimens if they also previously received neoadjuvant/adjuvant chemotherapy or chemoradiotherapy. The last treatment must have been administered > 3 weeks prior to initiation of therapy with sorafenib.
* Pathologic tissue must be available for immunohistochemistry (IHC) staining for phosphorylated extracellular signal-regulated kinase (pERK). Both patients with and without pERK staining are eligible for treatment. Submission of slides and IHC testing for pERK may be done during the course of therapy and are not required prior to protocol therapy.
* Age ≥ 18 years.
* Life expectancy > 3 months.
* Karnofsky performance status ≥ 60%.
* Patients must have the ability to comprehend and willingness to sign an informed consent document.
* At baseline, patients must have normal organ and marrow function as defined:

  * Adequate bone marrow, liver and renal function as assessed by the following:

    * Hemoglobin ≥ 9.0 g/dl
    * Absolute neutrophil count (ANC) ≥ 1,500/mm3
    * Platelet count ≥ 100,000/mm3
    * Total bilirubin ≤ 1.5 times ULN
    * ALT and AST ≤ 2.5 times the ULN ( < or = to 5 x ULN for patients with liver involvement)
    * Creatinine ≤ 1.5 times ULN

Exclusion Criteria:

* Patients who have not recovered from adverse events related to therapy administered > 3 weeks earlier. This does not include hemoglobin or other hematologic or laboratory criteria.
* Patients may not be receiving any other investigational agents.
* Prior therapy with sorafenib-related compounds or compounds of similar biologic or chemical components, including compounds targeting VEGF, VEGF-R or RAF kinase.
* Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, greater than New York Heart Association (NYHA) Class II congestive heart failure, unstable or new onset angina pectoris or myocardial infarction within the past six months, unstable arrhythmia, or psychiatric illness/social situation, e.g., severe schizophrenia, that would limit compliance with study requirements. Patients with chronic arrhythmias, such as paroxysmal atrial fibrillation or paroxysmal supraventricular tachycardia, are eligible.
* Uncontrolled hypertension, defined as systolic blood pressure > 150 mmHg or diastolic blood pressure > 90 mmHg, despite optimal medical management.
* Thrombotic or embolic event, including cerebrovascular accident or transient ischemic attack within the past six months. Patients with prior deep vein thromboses or pulmonary emboli on a stable anticoagulation regimen will be eligible for enrollment.
* Any factor that would significantly interfere with the inability to consume or absorb an oral medication, e.g. severe nausea/vomiting not controlled by an aggressive anti-emetic regimen, grade 3/4 dysphagia, extensive small bowel resection or active inflammatory bowel disease leading to chronic malabsorption. Patients with enteral feeding tubes are eligible as sorafenib can be crushed.
* Known human immunodeficiency virus (HIV) infection or chronic Hepatitis B or C infection.
* Patients with any other concurrent disease which, in the judgment of the investigator, would make the patient inappropriate for participation in the study.
* Patients who are taking St. John's wort or rifampin (as there may be drug-drug interactions with sorafenib.
* Patients with known brain metastases or meningeal carcinomatosis are excluded. Patients with neurological symptoms must undergo a CT scan/MRI of the brain to exclude brain metastasis.
* Pregnant women are excluded because sorafenib has the potential for teratogenic or abortifacient effects. Female patients must either not be of childbearing potential or must have a negative pregnancy test ≤ 7 days prior to treatment. Female patients are considered not of childbearing potential if they are surgically sterile (they have undergone a hysterectomy, bilateral tubal ligation or bilateral oophorectomy) or if they are post-menopausal. Men must use effective birth control if their partners are of child-bearing potential.
* No other malignancy is allowed except for adequately treated carcinoma in-situ of the cervix, superficial transitional cell carcinoma of the bladder or basal/squamous cell skin cancer. Other cancers are permissible if the patient has been disease free for ≥ 3 years.
* Pulmonary hemorrhage/bleeding event ≥ CTCAE Grade 2 within 4 weeks of first dose of study drug.
* Any other hemorrhage/bleeding event ≥ CTCAE Grade 3 within 4 weeks of first dose of study drug.
* Serious non-healing wound, ulcer, or bone fracture.
* Evidence or history of bleeding diathesis or coagulopathy.
* Major surgery, open biopsy or significant traumatic injury within 4 weeks of first study drug.
* Known or suspected allergy to sorafenib or any agent given in the course of this trial.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 35 (Actual)
Dates: Start 2009-06 (Actual); Primary Completion 2018-08 (Actual); Study Completion 2018-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: David Ilson, MD, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (1):
- Memorial Sloan Kettering Cancer Center, New York, New York, United States

REFERENCES:
- [Derived] Janjigian YY, Vakiani E, Ku GY, Herrera JM, Tang LH, Bouvier N, Viale A, Socci ND, Capanu M, Berger M, Ilson DH. Phase II Trial of Sorafenib in Patients with Chemotherapy Refractory Metastatic Esophageal and Gastroesophageal (GE) Junction Cancer. PLoS One. 2015 Aug 14;10(8):e0134731. doi: 10.1371/journal.pone.0134731. eCollection 2015. PMID 26275293
- See also: Memorial Sloan Kettering Cancer Center — http://www.mskcc.org

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Sorafenib
Started | 35
Completed | 34
Not Completed | 1
Not completed — Clinical Deterioration | 1

BASELINE CHARACTERISTICS:
Arm/Group | Sorafenib
Number analyzed (Participants) | 35
Age, Continuous [Median (Full Range); unit: years] | 62 [42 to 77]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4
  Male | 31
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1
  Not Hispanic or Latino | 34
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 3
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 31
  More than one race | 0
  Unknown or Not Reported | 1
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 35

OUTCOME MEASURES:

1. Primary Outcome: 2-month Progression-free Survival (PFS) of Sorafenib in Patients With Metastatic or Recurrent Esophageal and Gastroesophageal (GE) Junction Cancer.
Time Frame: 2 months
Measure: Count of Participants; unit: Participants
Arm/Group | Sorafenib
Number analyzed (Participants) | 35
Participants
  Progression Free | 20
  Progressed | 14
  Not evaluable | 1

2. Secondary Outcome: Overall Response Rate (Partial Response and Complete Response) of Sorafenib.
Description: Per Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.0) for target lesions and assessed by MRI: Complete Response (CR), Disappearance of all target lesions; Partial Response (PR), >=30% decrease in the sum of the longest diameter of target lesions; Overall Response (OR) = CR + PR.
Time Frame: after the first four weeks of therapy, at eight weeks, and every eight weeks thereafter, an average of 1 year
Measure: Count of Participants; unit: Participants
Arm/Group | Sorafenib
Number analyzed (Participants) | 35
Participants
  Disease Progression | 14
  Stable Disease | 19
  Complete Response | 1
  Not Evaluable | 1

3. Secondary Outcome: Number of Participants With Adverse Events
Time Frame: every week while on study
Measure: Count of Participants; unit: Participants
Arm/Group | Sorafenib
Number analyzed (Participants) | 35
Participants | 35

4. Secondary Outcome: Exploratory Analysis of Differential Response Between Squamous Cell Carcinoma and Adenocarcinoma.
Time Frame: 2 years
Population: Data were not collected
Arm/Group | Sorafenib
Number analyzed (Participants) | 0

5. Secondary Outcome: Percentage of Tumors With High Phosphorylated Extracellular Signal-regulated Kinase Expression
Time Frame: anytime prior to enrollment or during protocol therapy
Measure: Number; unit: % of tumors with high pERK expression
Arm/Group | Sorafenib
Number analyzed (Participants) | 35
% of tumors with high pERK expression | 65

ADVERSE EVENTS:
Time Frame: Up to 2 years
Arm/Group | Sorafenib
All-Cause Mortality (participants affected / at risk) | 35/35
Serious Adverse Events (participants affected / at risk) | 15/35
Other Adverse Events (participants affected / at risk) | 34/35
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Sorafenib (N=35)
Hyperbilirubinemia (Investigations) | 1
Hypercalcemia (Metabolism and nutrition disorders) | 1
Confusion (Psychiatric disorders) | 2
Constipation (Gastrointestinal disorders) | 1
Constitutional Symptoms, Other (General disorders) | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 1
Dehydration (Metabolism and nutrition disorders) | 4
Dry Mouth (Gastrointestinal disorders) | 1
Dysphagia (Gastrointestinal disorders) | 1
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1
Edema: viscera (General disorders) | 1
Fatigue (General disorders) | 2
Fever (General disorders) | 1
Fistula - GI, Esophagus (Gastrointestinal disorders) | 2
Hypertension (Vascular disorders) | 1
Pleural Infection (Infections and infestations) | 1
Motor neuropathy (Nervous system disorders) | 2
Pain - Chest Wall (Musculoskeletal and connective tissue disorders) | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1
Pain - Other (General disorders) | 1
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1
Renal/Genitourinary - Other (Renal and urinary disorders) | 1
Rigors/Chills (General disorders) | 1
Secondary malignancy (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Sinus Tachycardia (Cardiac disorders) | 1
Thrombosis/Thrombus/Embolism (Vascular disorders) | 1
Vomiting (Gastrointestinal disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Sorafenib (N=35)
Fatigue (General disorders) | 30
Diarrhea (Gastrointestinal disorders) | 18
Nausea (Gastrointestinal disorders) | 12
Dermatology/Skin - other (Skin and subcutaneous tissue disorders) | 10
Albumin, low (Metabolism and nutrition disorders) | 9
Anorexia (Metabolism and nutrition disorders) | 9
Hemoglobin/Anemia (Blood and lymphatic system disorders) | 9
Dry Skin (Skin and subcutaneous tissue disorders) | 8
Rash: hand-foot skin reaction (Skin and subcutaneous tissue disorders) | 8
Hyperglycemia (Metabolism and nutrition disorders) | 7
Vomiting (Gastrointestinal disorders) | 6
Constipation (Gastrointestinal disorders) | 5
Weight Loss (Investigations) | 5
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 4
Alopecia (Skin and subcutaneous tissue disorders) | 4
Mucositis (Gastrointestinal disorders) | 4
Sensory Neuropathy (Nervous system disorders) | 4
Platelets (Investigations) | 4
Rash/desquamation (Injury, poisoning and procedural complications) | 4
Hyponatremia (Metabolism and nutrition disorders) | 4
ALT/Alkaline phosphatase increased (Investigations) | 3
AST/Aspartate aminotransferase increased (Investigations) | 3
Alkaline Phosphatase (Investigations) | 3
Fever (General disorders) | 3
INR (Investigations) | 3
Lymphopenia (Investigations) | 3
Cough (Respiratory, thoracic and mediastinal disorders) | 2
Creatinine (Investigations) | 2
Hypertension (Vascular disorders) | 2
Leukocytes (Investigations) | 2
Lipase (Investigations) | 2
Pain - scalp (Skin and subcutaneous tissue disorders) | 2
Pain - skin (Skin and subcutaneous tissue disorders) | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2015-05-12): https://cdn.clinicaltrials.gov/large-docs/62/NCT00917462/Prot_SAP_000.pdf